CLINICAL TRIAL: NCT05725512
Title: Prednisolone Administration in Patients With Unexplained REcurrent MIscarriages, PREMI Trial
Brief Title: Prednisolone Administration in Patients With Unexplained REcurrent MIscarriages
Acronym: PREMI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Amsterdam University Medical Center (Other); Erasmus Medical Center (Other); Academisch Ziekenhuis Groningen (Other); Maastricht University Medical Center (Other); Isala (Other); Catharina Ziekenhuis Eindhoven (Other); Haaglanden Medical Centre (Other); Amphia Hospital (Other); Radboud University Medical Center (Other); Jeroen Bosch Ziekenhuis (Other); Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: Principal Investigator, E.E.L.O. Lashley, MD, Principle investigator, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LUMC-PREMI
Record Dates: First submitted 2023-01-19; First posted 2023-02-13 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Recurrent Miscarriage; Recurrent Pregnancy Loss; Habitual Abortion; Miscarriage; Fertility Disorders
Keywords: Recurrent pregnancy loss; Recurrent miscarriage; prednisolone
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: None of the personnel with patient contact will have knowledge to the patient's allocation to prednisolone or placebo group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prednisolone (Experimental): Prednisolone tablets (20 mg daily for 6 weeks, 10 mg daily for 1 week, 5 mg daily for 1 week)
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Identical placebo tablets for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Prednisolone — Prednisolone tablets (20 mg daily for 6 weeks, 10 mg daily for 1 week, 5 mg daily for 1 week) or identical placebo tablets for 8 weeks
  Arms: Prednisolone
Drug: Placebo — Placebo identical to prednisolone tablets
  Arms: Placebo

SUMMARY:
Recurrent miscarriages (RM) affects 3% of all fertile couples, but remains unexplained in most cases, limiting therapeutic options. Possibly the maternal immune system plays a role in recurrent miscarriage. Prednisolone suppresses the immune system and might enable development of normal pregnancy.

In this randomized controlled clinical trial the investigators will study the effect of prednisolone on the live birth rate in patients with RM. Secondary, the tolerability and safety for mother and child and the cost-effectiveness is investigated.

In the study one group of pregnant women with RM and gestational age <7 weeks will receive prednisolone, the other group will receive a placebo. Total use of the medicine during this study is 8 weeks, further care during the study is routinely antenatal care. Subjects will be asked to fill in 4 short questionnaires and will have contact with a research nurse at different time points to gain information on the course of the pregnancy and possible side effects.

Results of the study will be implemented in (inter) national guidelines, to effect everyday practice.

DETAILED DESCRIPTION:
Rationale:

Recurrent miscarriage (RM) is defined as 2 or more spontaneous miscarriages. It affects 3% of all fertile couples and in less than 50% an underlying cause may be identified. Thus far, none of the therapies tested in women with unexplained RM showed improvement of the live birth rate (LBR).

As the fetus is a semi-allograft, which escapes maternal immune rejection in normal pregnancy, many studies proposed the involvement of immunological mechanism in RM.

Glucocorticoids could have an effect on these mechanisms. Indeed, a recent meta-analysis has shown a beneficial effect on live birth rate for treatment with prednisolone therapy (RR 1.58, 95% CI 1.23-2.02). The included trials however were inadequately powered, differed in inclusion criteria or contained co-intervention with heparin and aspirin. In addition, most patients were selected based on the natural killer cell density in prior uterine biopsy, though this has not yet proven to be a valid biomarker.

Objectives:

To assess the effectiveness of prednisolone administration, as compared to placebo, on the LBR in an unselected population of women with unexplained RM.

Secondary, the effectiveness of prednisolone on the LBR in various subgroups, the tolerability and safety of prednisolone, the cost-effectiveness and the effect on immune cell levels is studied.

Main study parameters/endpoints:

Primary outcome: live birth rate Secondary outcome: miscarriage rate, ongoing pregnancy rate, adverse events (including side effects and pregnancy complications), decidual immune cell level and direct costs.

Trial design:

Randomized double-blind, placebo controlled multi-center clinical trial. Follow up period ends 3 months after delivery (12 months after randomization).

Trial population:

Women with unexplained recurrent miscarriage, including at least 2 miscarriages, aged 18- 39 years are recruited in a new pregnancy with AD <7 weeks from 10 participating centers in the Netherlands (Coordinating center Leiden University Medical Centre, LUMC).

Diagnosis unexplained recurrent miscarriages is based on latest ESHRE guideline.

Intervention:

After a complete diagnostic work-up, eligible women will be asked to collect a sample of menstrual blood. Patients are then randomized for prednisolone or placebo in a subsequent pregnancy. Women are randomly assigned in a 1:1 ratio to prednisolone tablets (20 mg daily for 6 weeks, 10 mg daily for 1 week, 5 mg daily for 1 week) or identical placebo tablets.

The participants will then receive prenatal visits according to standard care with their own treating physician. All patients will be asked to fill in questionnaires at randomization, and 3, 6 and 12 months after randomization. In a subgroup of patients participating in the LUMC and Radboud MC, additional analyses will be performed, aimed at elucidating the effect of prednisolone on level of different immune cell populations in miscarriage tissue or placenta.

Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks:

In the PREMI study the investigators will evaluate the effect of prednisolone on the live birth rate in patients with RM in a randomized, placebo-controlled trial. The risks and burden of participating in the trial are estimated as small. The risk of participation is the risk of prednisolone use; substantial evidence exists that prednisolone in this dosage and usage in first trimester is safe for mother and fetus.

Patients may however experience barriers for participation in this study, due to the possible assignment to the placebo-arm (with a possible nil effect on pregnancy outcome), as well as potential side effects. Considering the latter, in a previous feasibility trial no side effects were severe enough for women to stop taking medication. Moreover, to establish the most valid results as possible, there is no other solid manner to answer this research question than by conducting a well-designed double blinded placebo-controlled RCT.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Unexplained recurrent pregnancy loss: defined as the loss of ≥2 pregnancies, without any known cause for RM (parental chromosomal abnormalities, uterine anomalies, acquired or hereditary thrombophilia, endocrine diseases (such as hypothyroidism or diabetes)).
* The miscarriages include:

  * all consecutive or non-consecutive pregnancy losses before the 24th week of gestation verified by ultrasonography or uterine curettage and histology
  * non-visualized pregnancies (including biochemical pregnancy losses and/or resolved and treated pregnancies of unknown location), verified by positive urine or serum hCG Ectopic and molar pregnancies are not included
* Age 18 - 39 years at randomization (likelihood of miscarriages due to chromosomal aberrations is higher when age > 39 years. Such miscarriages are unlikely to be pre-vented by prednisolone therapy)
* Conception confirmed by urinary pregnancy test, with estimated gestational age ≤ 7weeks
* Willing and able to give informed consent in English or Dutch (IC)

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Any of the following diagnosis for the recurrent miscarriages

  * Antiphospholipid syndrome (lupus anticoagulant and/ or anticardiolipin anti-bodies and/or beta-2 glycoprotein [IgG or IgM)
  * Congenital uterine abnormalities (as assessed by 2D or 3d ultrasound, hys-terosonography, hysterosalpingogram or hysteroscopy)
  * Abnormal parental karyotype
* Instable or exacerbation of auto-immune diseases such as diabetes, thyroid disease, inflammatory bowel diseases or SLE
* Inability to conceive within 1 year of recruitment
* Current treatment with systemic prednisolone or other immune suppressive medication (for any indication)
* Previous enrolment in the PREMI trial
* Enrolment in any other trial that studies the effectiveness of an intervention on RM
* Contraindications to prednisolone use:

  * Known allergy for prednisolone
  * Acute bacterial infection or parasite infection
  * Active COVID infection
  * Systemic sclerosis
  * Ulcus ventriculi or ulcus duodeni in medical history
  * Obesity with BMI >40
* Some drugs are known to interact with Prednisolone, and thus women on the following drugs are not eligible to take part in the PREMI trial:

  * Enzyme inducers, such as carbamazepine, fenobarbital, fenytoïne and ri-fampicine
  * CYP3A inhibitors, such as Cobicistat or Ritonavir
  * Cyclosporine
  * Digoxin
  * Vaccination (with inactivated virus or bacteria) during prednisolone use is possibly less effective

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 490 (Estimated)
Dates: Start 2024-01-29 (Actual); Primary Completion 2026-07-29 (Estimated); Study Completion 2027-07-29 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | Within 24 months after eligibility
  Birth of a living child beyond 24 weeks

SECONDARY OUTCOMES:
Ongoing pregnancy | At +/- 12 weeks of pregnancy
  Fetal heartbeat on ultrasound scan at 12 weeks
Congenital abnormalities | At or short after birth, within 24 months after eligibility
  Number of children born with congenital deformity (such as cleft palate)
Gestational age | After birth, within 24 months after eligibility
  Gestational age measured in weeks after conception until delivery
Survival at 28 days of neonatal life | 28 days postpartum
  Is newborn still alive 28 days after birth
Adverse events | From start intervention until stop intervention (maximum of 7 weeks)
  Side effect of steroids (eg: insomnia, mood changes, indigestion)
Pregnancy complications | During pregnancy, maximum of 9 months
  Such as preeclampsia, pregnancy induced hypertension, HELLP and gestational diabetes
Direct and indirect costs | After intervention, after a maximum of 24 months
  Cost directly and undirectly related to intervention in comparrison to standard care
Anxiety and depression | Measurement at start of pregnancy (randomisation), 3, 6 and 12 months after start
  Anxiety and depression measured with questionnaire (HADS)
Quality of life (Health state) | Measurement at start of pregnancy (randomisation), 3, 6 and 12 months after start
  Quality of life measured through questionnaire (EQ-5D-5L) mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Birthweight | At birth, within 24 months after eligibility
  Measured in kilograms at time of birth
Productivity costs due to condition | 6 and 12 months after randomisation
  Productivity loss and costs measured through questionnaire (iPCQ)
Medical consumption | 6 and 12 months after randomisation
  Medical consumptoin expressed in e.g. number of visits measured through questionnaire (iMCQ)

OTHER OUTCOMES:
Level of immune cells post intervention | After miscarriage or delivery, within 24 months after eligibility
  level of uNK cells, regulatory T cells and CD14+/CD163+ macrophages in placenta or miscarriage tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Leiden University Medical Center, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Possibly various covariates among women with RM contribute to the effect of prednisolone on the live birth rate. To further study the effect of prednisolone in predefined subgroups we aim to conduct a individual participant data meta-analysis.
  These subgroups include groups defined on female age, number of previous miscarriages, antinuclear antibodies positivity and TPO antibodies positivity
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After results have been published in a manuscript.
Access Criteria: If informed consent of participants is available, individual data on above mentioned co-variates will be shared for IPD meta-analysis. Sharing will be done after publication and will be available up to 5 years after study has ended. Study protocol will be available too. Data will only be shared with researchers with a methodologically sound proposal directed to e.e.l.o.lashley@lumc.nl. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Bequet Y, van der Hoorn ML, Eikmans M, Van der Molen R, le Cessie S, van Geloven N, van den Akker-van Marle E, Vermeulen M, van den Berg M, de Bruin JP, Cantineau A, Huppelschoten D, Meuleman T, Mulders A, Al-Nasiry S, Teklenburg G, Verhoeve H, Visser J, van der Zanden M, Goddijn M, Lashley E. Effect of prednisolone on live birth rate in women with unexplained recurrent pregnancy loss: a study protocol for a double-blind, placebo-controlled, multicentre, randomised controlled trial (PREMI-study). BMJ Open. 2025 Jun 19;15(6):e096545. doi: 10.1136/bmjopen-2024-096545. PMID 40537239